CLINICAL TRIAL: NCT04012944
Title: A Prospective, Multi-Center, Open-Label, Single-Arm Clinical Trial Evaluating the Safety and Efficacy of the Cordella™ Pulmonary Artery Sensor System in New York Heart Association (NYHA) Class III Heart Failure Patients (SIRONA 2 Trial)
Brief Title: SIRONA 2 Trial Heart Failure NYHA Class III
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endotronix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ETX-HFS-PA-02
Record Dates: First submitted 2019-06-12; First posted 2019-07-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure NYHA Class III
Keywords: Heart Failure; Heart Diseases; Cardiovascular Disease
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cordella™ Pulmonary Artery Sensor System (Experimental): The Cordella PA Sensor System (CorPASS) is intended to measure, record, and transmit pulmonary artery pressure (PAP) data from NYHA Class III heart failure patients at home to clinicians for assessment and patient-centered heart failure management
  Interventions: Device: Cordella™ Pulmonary Artery Sensor System

INTERVENTIONS:
Device: Cordella™ Pulmonary Artery Sensor System — The Cordella PA Sensor System comprises seven subsystems that operate together to take daily Pulmonary Artery Pressure (PAP) readings at a patient's home and transmit the results to a care provider for evaluation.
  1. Cordella Sensor
  2. Cordella Delivery System
  3. myCordella Patient Reader
  4. Reader Dock
  5. Cordella Calibration Equipment (CalEQ)
  6. myCordella Hub
  7. Cordella Data Analysis Platform (CDAP).

SUMMARY:
This is a prospective, multi-center, open-label, single-arm CE-Mark trial to assess device safety and efficacy of the Cordella PA Sensor System in up to 75 New York Heart Association (NYHA) Class III Heart Failure patients who will receive the Cordella PA Sensor Implant.

DETAILED DESCRIPTION:
The study objectives are:

1. To establish that the Cordella PA Sensor can be safely delivered, deployed, and remain stable within the target pulmonary artery (PA) segment through 30 days post-implant.
2. To compare Cordella PA Sensor System pressure measurements with fluid-filled catheter PA pressure measurements obtained by standard right heart catheterization (RHC) at 90 days post implant.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent
2. Male or female, at least 18 years of age
3. Diagnosis of HF ≥ 6 months with either preserved or reduced left ventricular ejection fraction (LVEF) and NYHA Class III HF at the time of Screening
4. HF related hospitalization, HF treatment in a hospital day-care setting, or unplanned outpatient clinic HF visit within 12 months prior to consent and/or increase of N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) (or Brain Natriuretic Peptide (BNP)) at time of Screening defined as:

   1. Subjects with LVEF ≤ 40%: NT-proBNP ≥ 1000 pg/mL (or BNP ≥ 250 pg/mL).
   2. Subjects with LVEF > 40%: NT-proBNP ≥ 700 pg/mL (or BNP ≥ 175 pg/mL). Thresholds for NT-proBNP and BNP (for both LVEF ≤ 40% and LVEF > 40%) will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 25 kg/m2
5. Subjects must be receiving appropriate medical management of HF for 3 months prior to Screening and clinically stable for at least 1 month prior to study entry
6. Subjects who are physically able to hold the myCordella™ Patient Reader unit (approximate weight 600g) against the ventral thoracic surface for up to 2 minutes per day while in a seated position, as well as dock and undock the myCordella™ Patient Reader
7. Subjects with sufficient eyesight, hearing, and mental capacity to respond to the myCordella™ Patient Reader's audio/visual cues and operate the myCordella™ Patient Reader
8. Subject has sufficient Cellular and/or Wi- Fi Internet coverage at home
9. Subject agrees to return to the treating Investigator for all scheduled follow up visits and can return to the hospital for follow up

Exclusion Criteria:

1. Subjects with primary pulmonary hypertension
2. Subjects with an active infection at the Cordella PA Sensor Implant Visit
3. Subjects with history of pulmonary embolism or deep vein thrombosis
4. Subjects who have had a major cardiovascular event (e.g., myocardial infarction, stroke) within 2 months of the Screening Visit
5. Subjects whereby RHC is contraindicated
6. Implanted with a Cardiac Rhythm Management (CRM) Device (Internal Cardiac Defibrillator (ICD) or pacemaker) or Cardiac Resynchronization Therapy (CRT)-Pacemaker (CRT-P) or CRT-Defibrillator (CRT-D) less than 90 days prior to screening visit
7. Any major surgery within 30 days of the Sensor Implant Visit.
8. Subjects with a Glomerular Filtration Rate (GFR) <25 ml/min or who are on chronic renal dialysis
9. Specific liver enzymes [Aspartate Aminotransferase (AST) (SGOT), and Alanine Aminotransferase (ALT) (SGPT) >3 times the upper limit of normal
10. Received or are likely to receive an advanced therapy (e.g., mechanical circulatory support or lung or heart transplant) in the next 12 months
11. Subjects with congenital heart disease or mechanical/tissue right heart valve(s)
12. Subjects with known coagulation disorders
13. Subjects with a hypersensitivity or allergy to platelet aggregation inhibitors including aspirin, clopidogrel, prasugrel, and ticagrelor; or patients unable to take dual antiplatelet or anticoagulants for one- month post implant
14. Known history of life threatening allergy to contrast dye
15. Subjects who are pregnant or breastfeeding
16. Subjects who are unwilling or deemed by the Investigator to be unwilling to comply with the study protocol, or subjects with a history of non-compliance
17. Severe illness, other than heart disease, which would limit survival to <1 year
18. Subjects whose clinical condition, in the opinion of the Investigator, makes them an unsuitable candidate for the study
19. Subjects enrolled in another investigational trial with an active Treatment Arm
20. Subject who is in custody by order of an authority or a court of law
21. Unrepaired severe valvular disease
22. Subjects with an inferior vena cava (IVC) filter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Safety: Freedom from Adverse Events | 30 days
  To evaluate the primary safety endpoint: Freedom from AEs associated with use of the CorPASS through 30 days post Cordella PA Sensor implant, the number of subjects with and without any Adverse Device Events will be summarized.
Accuracy of Cordella PA Sensor System pressure measurements, compared to standard-of-care fluid-filled catheter PA pressure measurements obtained by standard Right Heart Catheterization (RHC) | 90 days
  System accuracy will be compared to the accuracy of standard-of-care commercial products that use fluid-filled invasive catheters to measure PA pressure at 90 days post implant visit.

SECONDARY OUTCOMES:
Frequency of Adverse Events | 30 days and 2 years
  Frequency of adverse events throughout the study
Device/system-related complications | 30 days and 2 years
  The rate of device/system-related complications will be assessed throughout the study
Pressure sensor failure rate | 30 days and 2 years
  Pressure sensor failure rate throughout the study
Accuracy using the Bland Altman Method | 90 days
  Accuracy of Cordella PA Sensor System pressure measurements, compared to standard-of-care fluid-filled catheter PA pressure measurements obtained by standard RHC using the Bland Altman method.
Accuracy of Cordella PA Sensor pressure measurements | 12 months
  Accuracy of Cordella PA Sensor System pressure measurements, compared to standard-of-care fluid-filled catheter PA pressure measurements obtained by standard RHC
Device Success | 90 days
  Percentage of device success as documented by ability of the System to successfully transmit collected PAP data to a secure database
Change in Pulmonary Artery (PA) pressure | 90 days and 2 years
  Change in PA pressure:
  1. Pre- and post-implant
  2. Before and after 6-Minute Walk Test
  3. Sitting vs supine PA pressure measurements
HF related hospitalizations, treatments in a hospital day-care setting, or urgent outpatient clinic visits. | 90 days and 2 years
  Frequency of HF hospitalizations, HF treatments in a hospital day-care setting, or urgent outpatient clinic HF visits.
Quality of Life measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) | 90 days and 2 years
  The Quality of Life KCCQ questionnaire is a measure of health-related quality of life. It is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life related to Heart Failure. Out of 23-items, 10 scores will be calculated: Physical Limitation, Symptom Stability, Symptom Frequency, Symptom Burden, Total Symptom Score, Self-Efficacy, Quality of Life, Social Limitation, Overall Summary Score, Clinical Summary Score .Presentation will be done by means of descriptive statistics including the absolute value and change from baseline by visit.
Adherence to regular myCordella™ Peripherals measurements measured as a percentage of subjects who adhere to regular myCordella™ Peripherals measurements | 90 days and 2 years
  Subjects will be instructed to perform daily measurements throughout the study. Subject compliance will be defined as at least 5 days of data collection/transmissions per week.
Heart Failure related medication changes | 90 days and 2 years
  Heart failure related medication change will be collected and summarized by visit presenting the percentage of subjects with and without any change in Heart Failure related medication
Functional Status Change as measured by New York Heart Association (NYHA) functional classification | 90 days and 2 years
  The NYHA functional classification categorizes the extent of heart failure by placing subjects in one of four (I, II, III, IV) categories based on how much they are limited during physical activity and symptoms of shortness of breath and/or angina. Shifts in NYHA functional classification from baseline over all post-baseline visits will be presented.
Functional Status Change as measured by 6-Minute Walk Test | 90 days and 2 years
  Subjects complete a six (6) minute walk test at the study visits described in the study protocol. Total distance walked (meters) will be collected and analyzed by means of descriptive statistics including the absolute value and change from baseline by visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sauerland, Study Director — Endotronix, Inc.
Locations (7):
- Belgium (2):
  - Cardivascular Center OLV Aalst, Aalst
  - Ziekenhuis- Oost Limburg, Genk
- Germany (3):
  - Uniklinik Köln, Klinik III für Innere Medizin Herzzentrum der Universität zu Köln, Cologne
  - Universitätsklinikum Giessen und Marburg GmbH, Standort Giessen Medizinische Klinik I, Abteilung Kardiologie und Angiologie, Giessen
  - Klinik für Kardiologie und Angiologie/ Studienambulanz Medizinische Hochschule Hannover (MHH), Hanover
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - University Hospital Galway, Dublin